CLINICAL TRIAL: NCT03577548
Title: Influence of Main Psychological and Social Factors on Primary Headaches
Acronym: CEPHAPSY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/290
Record Dates: First submitted 2018-03-26; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Auto- questionnaires — 10 auto-questionnaires are submitted to the patient during his/her consultation (which is part of the standard care).

SUMMARY:
This study aims to describe the psychological and social characteristics of patients suffering from primary headache and monitored in Neurology department of Besançon University Hospital

DETAILED DESCRIPTION:
The aim of our study is to describe the psychological patterns in a population of patients suffering of episodic migraine or chronic migraine with and without medication overuse and the level of disability.

Data about migraine characteristics will be obtained using a standardized questionnaire.

Socio-demographic data will be obtained for all patients including gender, age, educational level and professional status.

A booklet of 10 self-administered questionnaires will permit to measure psychological factors such as depression, anxiety, alexithymia...

ELIGIBILITY:
Inclusion Criteria:

* Patients from 25 to 60 ans y.o suffering from primary headache and monitored in the Neurology department of Besançon University Hospital

Exclusion Criteria:

* Patients with former or current psychic troubles

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All subjects are suffering from primary headache and come for come for a specialized consultation in the Neurology department of Besançon University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05-02 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Descriptive analysis of socio-demographic questionnaire | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
Descriptive analysis of Short Form 36 (SF 36) Health Survey | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
  This questionnaire asseses quality of life.
Descriptive analysis of General Health Questionnaire 12 | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
  Ranges for this questionnaire: 0 - 1 : no psychological distress / 2 - 3 : psychological problems / 4 - 48 : suspicion of mental illness.
Descriptive analysis of Cungi test | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
  Ranges for this questionnaire: 12 - 19 : very low level of stress / 20 - 30 : low level of stress / 31 - 45 : high level of stress / > 45 : very high level of stress.
Descriptive analysis of State-Trait Anxiety Inventory Y-A | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
  Ranges for this questionnaire (current anxiety): < 36 : very low / 36 à 45 : low / 46 à 55 : medium / 56 à 65 : high / > 65 : very high.
Descriptive analysis of State-Trait Anxiety Inventory Y-B | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
  Ranges for this questionnaire (general anxiety): < 36 : very low / 36 à 45 : low / 46 à 55 : medium / 56 à 65 : high / > 65 : very high.
Descriptive analysis of Beck Depression Inventory | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
  Ranges for this questionnaire: 0 - 4 : no depression / 5 - 7 : mild depression / 8 - 15 : moderate depression / > 15 : severe depression.
Descriptive analysis of Social Support Questionnaire 6 | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
  This questionnaire assesses satisfaction upon social support.
Descriptive analysis of Toronto Alexithymia Scale 20 | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
  Three levels for alexythimia: < 44 : non-alexithymia / 44 à 55 : possible alexithymia / > 55 : alexithymia.
Descriptive analysis of Bartholomew Relationship Scales Questionnaire | Day 1
  Composite outcome assessed with 10 questionnaires are submitted to the patients and all their results are combined in order to identify psychological and social characteristics of the patients:
  Quantitative variables will be mean, standard deviation, median and minimal/maximal values. Qualitative variables will be described by frequency and proportion of each class.
  Four levels for this questionnaire: Secure, Preoccupied, Dismissing and Fearful.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belot RA, Bouteloup M, Bonnet M, Parmentier AL, Magnin E, Mauny F, Vuillier F. Evaluation of Attachment Style and Social Support in Patients With Severe Migraine. Applications in Doctor-Patient Relationships and Treatment Adherence. Front Neurol. 2021 Jul 12;12:706639. doi: 10.3389/fneur.2021.706639. eCollection 2021. PMID 34322089
- [Derived] Bouteloup M, Belot RA, Noiret N, Sylvestre G, Bertoux M, Magnin E, Vuillier F. Social and emotional cognition in patients with severe migraine consulting in a tertiary headache center: A preliminary study. Rev Neurol (Paris). 2021 Oct;177(8):995-1000. doi: 10.1016/j.neurol.2020.09.013. Epub 2021 Jan 13. PMID 33454126